CLINICAL TRIAL: NCT03276481
Title: Prospective Evaluation of Gustatory Function (Taste) In Patients Undergoing Autologous Hematopoietic Cell Transplantation for Multiple Myeloma
Brief Title: Prospective Evaluation of Taste Function In Multiple Myeloma Patients Undergoing Autologous Hematopoietic Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-404
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
Keywords: melphalan; stem cell transplantation; 17-404; hematopoietic cell transplantation; HCT
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Myeloma: Participants with multiple myeloma undergoing autologous hematopoietic cell transplantation (HCT) after a high dose melphalan conditioning regimen
  Interventions: Diagnostic Test: Oral microbiota assessment; Diagnostic Test: Comprehensive chemical gustometry; Diagnostic Test: Measurement of salivary flow; Behavioral: Surveys assessing taste disturbances

INTERVENTIONS:
Diagnostic Test: Oral microbiota assessment — Whole mouth microbiota will be assessed by having participants swish in their mouth 10 ml of sterile water for 30 sec and then expectorate in a sterile container. Specimens will be immediately placed on wet ice and transferred to the laboratory for processing or for storage at -80° C until they are ready to be prepared for sequencing.
Diagnostic Test: Comprehensive chemical gustometry — Chemical gustometry assessments will be performed by a trained clinician on the study team, including a Registered Dietitian, Physician's Assistant, or Research Nurse. The test solutions and gradients will be formulated in house using sterile water and the following constituents: Sweet taste; 0.05, 0.1, and 0.2 g/ml sucrose, sour taste; 0.05, 0.09, and 0.165 g/ml citric acid, salty taste; 0.016, 0.04, and 0.1 g/ml NaCl and bitter taste; 0.0004, 0.0009, and 0.0024g/ml quinine-HCl. Umami will be tested with MSG at 25, 50, and 75 mM.
Diagnostic Test: Measurement of salivary flow — Both stimulated and un-stimulated salivation will be assessed by saliva collection in pre-weighed plastic containers. Participants will be seated with their back at a 90 degree angle and asked to swallow everything in their mouth. They will then be asked not to swallow and spit the accumulated saliva in the plastic container every 30 seconds for two minutes (unstimulated flow). For measurement of stimulated saliva, we will follow the same procedure except that after the initial swallow, participants will have their tongue swabbed twice with a cotton swab dipped in ascorbic acid solution or lemon juice.
Behavioral: Surveys assessing taste disturbances — Surveys will be administered and examine taste disturbances pre and post HCT.

SUMMARY:
The purpose of this study is to study taste disturbances on patients with myeloma who received high dose melphalan.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or above with diagnosis of multiple myeloma (myeloma is almost unheard of in patients less than 21 years of age).
* Scheduled to receive conditioning chemotherapy with melphalan followed by upfront or salvage autologous peripheral blood hematopoietic stem cell transplantation
* English or Spanish speaking
* Calculated creatinine clearance > 40 mL/min

Exclusion Criteria:

* Prior head and neck radiation.
* Severe periodontal infection. Poor oral hygiene and dentition as determined by pre HCT dental assessment.
* Pregnancy
* Patients with pre-existing moderate-severe dysgeusia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be identified by the Adult Bone Marrow Transplant team. They are usually identified in clinic when a treatment plan that includes conditioning chemotherapy has been scheduled.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of comprehensive chemical gustometry in participants with multiple myeloma undergoing autologous HCT | Change from baseline assessment up to 100 days
  The primary objective of this protocol is to evaluate the feasibility of comprehensive chemical gustometry in participants with MM undergoing autologous HCT. Chemical gustometry will be evaluated at baseline and on days -1, 7, 14, 30 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org